CLINICAL TRIAL: NCT00082069
Title: Safety and Immunogenicity Study of an Intranasal Shigella Flexneri 2a Invaplex 50 Vaccine
Brief Title: Invaplex 50 Vaccine Dose-Ranging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NMRC 2003.0006; WRAIR 1085 (Other: WRAIR); HSRRB A-12528 (Other: USAMRMC)
Record Dates: First submitted 2004-04-28; First posted 2004-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Diarrhea
Keywords: Shigella; diarrhea
MeSH Terms: conditions — Diarrhea; Dysentery, Bacillary

INTERVENTIONS:
Biological: Shigella flexneri 2a Invaplex 50

SUMMARY:
The vaccine is given as a nose spray. Volunteers will receive a 3-dose vaccination with doses spaced two weeks apart. Volunteers will be assigned to a vaccination group based on their order of enrollment with consideration of their availability to complete the necessary vaccinations and follow-up visits.

DETAILED DESCRIPTION:
This is an open-labeled dose escalating trial in which a total of 32 subjects (minimum of 24 allowable) will receive one of four intranasal Invaplex 50 vaccine doses according to the following chart:

Test articles/dose

Group / N* / Invaplex 50

A / 8 / 10 micrograms

B / 8 / 50 micrograms

C / 8 / 240 micrograms

D / 8 / 480 micrograms

*minimum of 6 volunteers/group

An interval no less than 7 days following the third (and final) dose (total of 35 days between initial dose at the lower dose level and the next initial dose at the next higher dose level) will separate volunteer groups receiving different doses. All volunteers will receive three immunizations. The first dosing time point is Day 0, the second is Day 14 (+- one day), and the third is Day 28 (+- 2 days). Blood and stool specimens will be collected at intervals to examine systemic and mucosal vaccine antigen-specific immune responses. Vaccine safety will be actively monitored during vaccination and for 28 days following the third vaccination dose.

ELIGIBILITY:
Inclusion Criteria:

* Be in very good health.

Exclusion Criteria:

* Smoker, or have stopped smoking less than one year ago
* Pregnant
* History of chronic illnesses, such as: asthma, chronic sinusitis, or chronic seasonal allergies (such as hay fever)
* Received a vaccination for Shigella or exposure to Shigella bacteria in a research study or through work in a laboratory
* Positive for HIV, hepatitis B, and hepatitis C by blood test
* Using anti-diarrheal, anti-constipation, or antacid medications on a regular basis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2004-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Safety
Mucosal immune response
Systemic immune response

CONTACTS AND LOCATIONS:
Overall Officials: David Tribble, MD, PhD, Principal Investigator — Naval Medical Research Center
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

REFERENCES:
- [Derived] Tribble D, Kaminski R, Cantrell J, Nelson M, Porter C, Baqar S, Williams C, Arora R, Saunders J, Ananthakrishnan M, Sanders J, Zaucha G, Turbyfill R, Oaks E. Safety and immunogenicity of a Shigella flexneri 2a Invaplex 50 intranasal vaccine in adult volunteers. Vaccine. 2010 Aug 23;28(37):6076-85. doi: 10.1016/j.vaccine.2010.06.086. Epub 2010 Jul 7. PMID 20619378